CLINICAL TRIAL: NCT03514056
Title: Frequency of Fibromyalgia in Behcet Disease in Province Bursa
Brief Title: Frequency of Fibromyalgia in Behcet Disease
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Koray Ayar, Assistant Professor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2018/03-14
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Fibromyalgia; Behcet Syndrome
Keywords: Fibromyalgia; Behcet Disease; Trigger points
MeSH Terms: conditions — Fibromyalgia; Behcet Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: group Behcet
  Interventions: Diagnostic Test: group 1:Patients diagnosed with Behcet disease
- 2: group fibromyalgia
  Interventions: Diagnostic Test: group 2: Patient diagnosed with fibromyalgia without Behcet disease

INTERVENTIONS:
Diagnostic Test: group 1:Patients diagnosed with Behcet disease — Frequency and severity of fibromyalgia will be investigated in patient diagnosed with Behcet disease
  Groups: 1
Diagnostic Test: group 2: Patient diagnosed with fibromyalgia without Behcet disease — Severity of fibromyalgia will be investigated in patient diagnosed with fibromyalgia
  Groups: 2

SUMMARY:
In various studies, the incidence of fibromyalgia in Behçet's patients is widely distributed. It was aimed to investigate the frequency and severity of fibromyalgia in Behcet disease in province Bursa.

DETAILED DESCRIPTION:
There are few studies in the literature investigating the frequency of fibromyalgia in Behçet's disease. In various studies, the incidence of fibromyalgia in Behçet's disease was 5.7% -37.1%, which is widely distributed. There are no studies in literature comparing disease severity and pain thresholds at trigger points in fibromyalgia with and without Behcet's disease. In this study, it was aimed to investigate the frequency of fibromyalgia in Behcet's disease according to the criteria defined by the American Colloge of Rheuatology in 2010 and updated in 2013. It was also aimed to compare the severity of disease in fibromyalgia with and without Behcet's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Behcet disease according to international study group criteria
* Patients diagnosed with fibromyalgia according to classification criteria that were defined by the American Collage of Rheumatology in 2010 and updated in 2013
* Patients older than 18
* Patients younger than 75

Exclusion Criteria:

* Participants which were previously diagnosed with diabetes mellitus
* Participants which were previously diagnosed with chronic renal failure
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of participants who are between age 18-75, not pregnant and who were not diagnosed previously with diabetes mellitus or chronic renal failure
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
fibromyalgia 2013 criteria | Six months
  Fibromyalgia 2013 criteria were derived from the 10-item symptom score from the Symptom Impact Questionnaire (SIQR) symptoms and the 28-area pain location inventory (PLI). If the patients PLI score is above 17 (range 0-28) and an SIQR symptom score is above 21 (range 0-50), the participant will be diagnosed with fibromyalgia

SECONDARY OUTCOMES:
Fibromyalgia impact questionnaire | Six days
  The fibromyalgia impact questionnaire (FIQ) has 21 individual questions . All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'. In the FIQ, all questions are framed in the context of the past 7 days. The total maximal score of the FIQ is 100.
Pain thresholds | Six months
  Pain thresholds will be recorded by applying pressure to the 28 sensitive points until the participants demonstrate pain. Manual algometry device will be used to measure the pain threshold.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Education and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided